CLINICAL TRIAL: NCT05803369
Title: Regulating Together: Randomized Controlled Trial Examining Predictors, Facilitators, and Barriers to Treatment Success in Emotion Dysregulation and Autism Spectrum Disorder (ASD)
Brief Title: DOD Regulating Together Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-22-1-0168; CDMRP-AR210169 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Autism Spectrum Disorder; Emotion Regulation
Keywords: Regulating Together
MeSH Terms: conditions — Autism Spectrum Disorder; Emotional Regulation | interventions — Schools

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regulating Together (RT) (Experimental): Participants will receive Regulating Together -the emotion dysregulation intervention
  Interventions: Behavioral: Regulating Together (RT)
- Achieving Independence and Mastery in School (AIMS) (Active Comparator): Participants will receive AIMS, the academic functioning/organizational skill intervention.
  Interventions: Behavioral: Achieving Independence and Mastery in School (AIMS)

INTERVENTIONS:
Behavioral: Regulating Together (RT) — Regulating Together is an intensive outpatient group treatment targeting emotion dysregulation. It engages both caregivers and children and utilizes evidence-based intervention techniques including cognitive behavioral therapy (CBT), visuals, reinforcements, and scaffolding, and newer interventions such as mindfulness and acceptance-based therapy.
  Arms: Regulating Together (RT)
Behavioral: Achieving Independence and Mastery in School (AIMS) — AIMS is a school-based program developed to help students with social-communication challenges (such as autism spectrum disorder) achieve academic success. It is well-established and has been used with autistic youth, both in schools and in outpatient settings.
  Arms: Achieving Independence and Mastery in School (AIMS)

SUMMARY:
Our long-term goal is to validate Regulating Together (emotion regulation intervention) and improve psychosocial outcomes for youth with autism spectrum disorder and emotion dysregulation.

DETAILED DESCRIPTION:
144 children ages 8-12 years old with autism spectrum disorder will be enrolled in the study and randomized to Regulating Together (RT) or Achieving Independence and Mastery in School (AIMS) groups. Participants will complete assessments at five time points: Screen (T1) Week 0 - where they will complete consent; Baseline (T2); Week 7: Post Active Treatment (includes semi-structured interviews) (T3); Week 16: Post Generalization (T4); Week 29: Final outcome visit (T5). Participants will receive 5 weeks of intervention, twice per week, following the T2 visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder (ASD)
* A Full Scale IQ score of 65 or greater on the Weschler Abbreviated Scale Intelligence (WASI-II) or other previous Weschler IQ test
* Concern of emotion dysregulation (ED) as measured by a score of 6 or greater on the Emotion Dysregulation Inventory-Reactivity (EDI-R).
* Caregivers and child are fluent in speaking English
* Child functional verbal communication, confirmed via appropriateness for an Autism Diagnostic Observation Schedule (ADOS-2) Module 3.
* Family willing to keep prescribed medication and outside interventions stable
* willing to participate in twice weekly 90-minute sessions of either Regulating Together (RT) or Achieving Independence and Mastery in School (AIMS).
* The guardian must provide written informed consent on behalf of the participant and the participants ages 11-12 years old must provide written informed assent to participate.

Exclusion Criteria:

* Initiation of new psychosocial intervention within 30 days prior to randomization/first day of treatment.
* any physical aggression toward other children outside the home in the past 2 weeks that resulted in serious injury
* Presence of comorbid major neuropsychiatric illness warranting other treatment approaches.
* Presence of any major sensory impairment that would limit participating in the material including blindness or uncorrected hearing loss

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Emotion Dysregulation Inventory- Reactivity | Through study completion, about 29 weeks
  13-item parent report measure that captures negative emotional responses and Dysphoria characterized by increased negative affect and lack of motivation. Higher scores mean higher emotional reactivity.

SECONDARY OUTCOMES:
Children's Organizational Skills Scale (COSS) | Through study completion, about 29 weeks
  Used to measure outcomes from AIMS intervention. It is a rating scale completed by parents and teachers which yields three factors measuring Organized Actions, Task Planning, and Memory and Materials Management. Higher scores mean higher organizational skills.
Daily Phone Diary | Through study completion, about 29 weeks
  Phone interview administered by staff that documents Frequency and Intensity of Behavioral and Emotional Outbursts over a 2 day period.
Inpatient Hospitalization Rates | during the 6 months prior to enrollment in the study and during the 6 months after completion of the individualized consult
  chart review and caregiver report for any psychiatric hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Shaffer, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] McKinney WS, Tadevich LJ, Schmitt LM, Horn PS, Ruberg JR, White SW, Reisinger DL, Burkett KW, Sarawgi S, Kang S, Shaffer RC. Study protocol for a randomized controlled trial of Regulating Together (RT), a group therapy for emotion dysregulation in school-age autistic youth and their caregivers. BMC Psychol. 2025 Apr 24;13(1):436. doi: 10.1186/s40359-025-02737-6. PMID 40275407